CLINICAL TRIAL: NCT02639221
Title: PXT002331 A Phase I, Double Blind, Placebo Controlled, First in Human, Single and Multiple Ascending Oral Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Male and Female Subjects
Brief Title: A Phase I, Double Blind, Placebo Controlled, First in Human, Single and Multiple Ascending Oral Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prexton Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: PXT-CL15-001
Record Dates: First submitted 2015-12-17; First posted 2015-12-24 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- PXT002331 (Experimental)
  Interventions: Drug: PXT002331
- Placebo (Placebo Comparator)
  Interventions: Drug: PXT002331

INTERVENTIONS:
Drug: PXT002331

SUMMARY:
The principal aim of this study is to obtain safety and tolerability data when PXT002331 is administered orally as single and multiple doses to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be; 1.1. males or females of non childbearing potential 1.2. For females, non childbearing potential is defined as follows:

   * permanently sterile following hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or confirmed tubal occlusion (not tubal ligation)
   * postmenopausal, defined as at least 1 year post cessation of menses (without an alternative medical cause) 1.3. of any ethnic origin 1.4. between 18 and 60 years of age, inclusive
2. Subjects will have a 2.1. body mass index (BMI) between 18.0 kg/m2 and 32.0 kg/m2, inclusive 2.2. body weight between 50 kg and 100 kg, inclusive
3. Subjects will be in good health, as determined by; 3.1. medical history 3.2. physical examination 3.3. vital signs assessment 3.4. 12 lead ECG and 24 hour Holter Monitoring 3.5. clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia is not acceptable)
4. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Serious Adverse Events | 16 days
Number of clinically relevant signs or symptoms | 16 days

CONTACTS AND LOCATIONS:
Locations (1):
- United Kingdom, United Kingdom, United Kingdom